CLINICAL TRIAL: NCT07383272
Title: We Need to F.E.E.D.: Facilitating Enteral Education for Discharge - Improving the Quality of Discharge for Pediatric Patients With Enteral Tubes
Brief Title: We Need to FEED: Facilitating Enteral Education for Discharge
Acronym: WeNeed2FEED
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Illinois at Chicago (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Supportive Care
Other Study IDs: STUDY2025-0139; NASPGHAN contract award 39608 (Other Grant/Funding Number: NASPGHAN Foundation/APGNN Susan Moyer Nursing Research Grant)
Record Dates: First submitted 2025-02-21; First posted 2026-02-03 (Actual); Last update posted 2026-02-03 (Actual); Status verified 2026-01

CONDITIONS: Enteral Nutrition Feeding
Keywords: education; feeding tube; g tube; ng tube; gj tube; parent education; pediatrics; patient education
MeSH Terms: interventions — Early Intervention, Educational

STUDY DESIGN:
Intervention Model Description: Investigators will have pre and post test for both the control and intervention group. the pretest will be administered before the education intervention is applied. This will be a quasi-experiemental design.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Usual Care (No Intervention): Usual care group will receive usual care/education provided at UI health on feeding tubes.
- Education (Experimental): Education Intervention provided to the intervention group. Intervention will include education handbook, onsite or via zoom education of g tube, question and answer.
  Interventions: Other: Education Intervention

INTERVENTIONS:
Other: Education Intervention — Education on feeding tubes, booklet, inperson or via zoom education to parents of pediatric patients with newly placed feeding tube ( G-tube, GJ-tube, NG tube). Education on supply company and how to get supplies. The need for back up feeding tube etc. Size of patient feeding tube.
  Arms: Education

SUMMARY:
Aim: We need to FEED (Facilitating Enteral Education for Discharge) project aims to streamline and enhance the discharge process for pediatric patients with enteral nutrition (including G-tubes, J-tubes, GJ-tubes, and NG-tubes) and ultimately create enteral discharge protocol. The aim of the study is to describe the effectiveness of the discharge education program for children with enteral tubes on caregiver knowledge and determine the impact of the program on unplanned ER, Urgent care or clinic visits. By ensuring that all necessary supplies, orders, and follow-up appointments are in place prior to discharge, and by providing comprehensive education and support to parents, the project seeks to improve patient outcomes, reduce healthcare utilization, enhance coordination and communication among healthcare providers.

DETAILED DESCRIPTION:
Objectives and Hypothesis Objective: The primary objective of the FEED project is to enhance the discharge process for pediatric patients with enteral nutrition, ensuring adequate education, all necessary supplies, orders, follow-up appointments are in place, thereby improving patient outcomes and reducing healthcare utilization. The secondary objective of the FEED project is to create a standardized enteral discharge protocol. Tertiary goal includes ensuring video swallow studies are completed inpatient to expedite feeding therapy

Hypothesis: The implementation of a structured discharge process for enteral nutrition patients will result in:

1. Reduced number of calls to the NICU, PEDS, PICU, outpatient pediatric and GI departments.
2. Decreased number of unplanned visits to emergency room, urgent care, clinic visits related to enteral nutrition issues.
3. Improved parent confidence and competence in managing enteral nutrition at home.
4. Streamlined access to early intervention and speech therapy services.
5. Enhanced coordination and communication among healthcare providers. Needs Assessment: Gastrostomy tubes (G-tubes) are commonly utilized to facilitate nutrition, hydration, and medication administration in children who have chronic inadequate oral intake due to conditions such as dysphagia, neurological disorders, chronic illnesses, oncologic problems, and other clinical conditions leading to malnutrition. Although G-tube placement is generally safe and frequently performed among pediatric patients, complications such as tube blockage, infection, and over granulation tissue are reported at varying frequencies. Home care plays a significant role in the occurrence of these common, minor, and preventable complications.

Research indicates that families often face challenges in managing home care for children with G-tubes due to insufficient knowledge and inadequate discharge support from healthcare professionals. Many families report that they have not been adequately informed by healthcare providers during discharge, leading to difficulties in providing correct care and disease management. The primary issues in home care include feelings of guilt due to the necessity of tube feeding, difficulties in daily care arising from tube-related complications, and fear of potential complications associated with enteral nutrition. The long-term nature of enteral feeding with G-tubes further increases the burden of care on families.

The American Society for Parenteral and Enteral Nutrition (ASPEN) emphasizes the importance of providing discharge education to patients with chronic illnesses and specific nutritional needs and maintaining safe home nutrition. Implementing a standardized, evidence-based discharge education protocol is expected to improve treatment outcomes, increase caregiver knowledge, and reduce the burden of care and anxiety levels.

The FEED (Facilitating Enteral Education for Discharge) project addresses these identified needs by streamlining the discharge process for pediatric patients with enteral nutrition. The project aims to ensure that all necessary supplies, orders, and follow-up appointments are in place prior to discharge. It also focuses on providing comprehensive education and support to parents, thereby improving patient outcomes, reducing healthcare utilization, and enhancing coordination and communication among healthcare providers. By addressing these key areas, the FEED project aims to improve the overall care for pediatric patients with enteral nutrition, ultimately enhancing patient outcomes and reducing the healthcare burden on families.

ELIGIBILITY:
Inclusion Criteria:

* Patients must be within the age range of 0 to 17 years.
* Patients who have recently had an enteral feeding tube placed (G-tube, J-tube, GJ-tube, or NG-tube).
* The patient must be hospitalized at the time of the study and scheduled for discharge within the study period (before discharge).
* A legal guardian must be available to participate in the study, complete questionnaires, and engage in the educational sessions.
* Both the pediatric patient and their caregiver must be willing to participate in the study, including completing surveys and receiving educational materials.

Exclusion Criteria:

* Patients who have had an enteral tube (G-tube, J-tube, GJ-tube, or NG-tube) for more than a short period (e.g., those who have had tubes in place for more than 3 months) may be excluded, as the study is focused on newly placed feeding tubes.
* Patients aged 18 years or older are excluded from the study, as the project targets pediatric patients specifically.
* If the caregiver (or the child, where applicable) has significant cognitive or language barriers that would prevent them from understanding the educational content or completing the surveys, they may be excluded.
* Families who do not speak English may be excluded.
* Patients with significant comorbidities or unstable clinical conditions that would make participation in the discharge education protocol impractical will be excluded. This includes, but is not limited to, patients with severe respiratory failure requiring nitric oxide therapy, hemodynamic instability requiring blood pressure medications (e.g., vasopressors), or other acute medical conditions requiring active intensive care. Patients who are stable and preparing for discharge, even after a prolonged NICU or PICU stay, will not be excluded.
* Only legal guardian can enroll child.
* Patients whose caregivers are unable or unwilling to adhere to study protocols (e.g., participating in follow-up assessments or completing questionnaires) may be excluded to ensure consistency and reliable data collection.

Max Age: 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 20 (Estimated)
Dates: Start 2026-02-01 (Estimated); Primary Completion 2027-03-31 (Estimated); Study Completion 2028-05-01 (Estimated)

PRIMARY OUTCOMES:
Families Enteral tube knowledge:Change in Enteral Tube Knowledge Score From Baseline and post hospital discharge | Baseline (while hospitalized prior to initial educational session in the hospital) and after discharge ( up to 3 months)
  Enteral tube knowledge will be measured using a enteral nutrition knowledge likert scale survey at baseline (hospitalized: at time of feeding tube placement and post discharge. Knowledge scores will be compared between the intervention group (FEED Program) and the control group (usual care).
Number of Unplanned Healthcare Visits Related to Enteral Tube Issues | post hospital discharge-through study completion, an average 1 year
  The number of unplanned healthcare visits (emergency department visits, urgent care visits, and unplanned outpatient visits) related to enteral tube complications will be tracked. Data will be compared between the intervention group (FEED Program) and the control group (usual care) to evaluate the program's impact on reducing unplanned healthcare utilization.

CONTACTS AND LOCATIONS:
Overall Officials: Kiranmai Gorla, MD, Study Chair — UI Health
Locations (1):
- University of Illinois at Chicago (UI Health), Chicago, Illinois, United States

IPD SHARING:
Plan to Share IPD: Undecided
Individual Participant Data (IPD) Sharing Statement
  1. Considerations for Data Sharing
  At this time, a final decision has not been made regarding the sharing of Individual Participant Data (IPD). Several factors influence whether IPD will be shared, including:
  Confidentiality and Privacy Concerns: Given the sensitive nature of patient and caregiver data, ensuring that all shared data is fully de-identified while maintaining participant privacy is a priority. Additional steps may be required to protect anonymity, which could impact data availability.
  Regulatory and Institutional Policies: Data-sharing decisions must align with institutional policies, HIPAA regulations, and ethical standards. Institutional Review Board (IRB) requirements may place restrictions on data distribution.
  Feasibility of Secure Data Sharing: Establishing a HIPAA-compliant, secure data-sharing platform requires resources. The availability of these resources will determine whether data can be shared responsibly

REFERENCES:
- [Background] Goldberg E., Kaye R., Yaworski J., Liacouras C. (2005). Gastrostomy tubes: facts, fallacies, fistulas and false tracts. Gastroenterology Nursing, 28(6): 485-493.
- [Background] DeLegge, M (2019). Gastrostomy Tubes: Complications and their management, Up To Date DeLegge, M (2019). Gastrostomy Tubes: Placement and routine care, Up To Date
- [Background] Crawley-Coha, T. (2004). A practical guide for the management of pediatric gastrostomy tubes based on 14 years' experience. Journal of Wound Ostomy and Continence Nursing, July/Aug 193-200.